CLINICAL TRIAL: NCT06346405
Title: Central Serous Chorioretinopathy and Micropulse Laser Treatment: Evaluation of Morphological and Functional Recovery
Brief Title: Central Serous Chorioretinopathy and Micropulse Laser Treatment
Acronym: LEVEO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Savastano Maria Cristina, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 10
Record Dates: First submitted 2024-03-05; First posted 2024-04-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Subthreshold Micropulse Laser Treatment — Subthreshold micropulse laser treatment consists in 33 spots of 100 microns, distance among each spot of 2.50 microns, duration of 200 sec, power of 250 milliwatt (mW) duty cycle 5%.

SUMMARY:
To evaluate choroidal and choriocapillaris changes in patients with central serous chorioretinopathy, undergone sub threshold micropulse laser treatment, following any improvement with conservative therapy with Acetazolamide and/or Eplerenone

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of central serous chorioretinopathy (CSC) with no response to conservative therapy, consisted in Acetazolamide and Eplerenone after six months.
* Foveal serous retinal detachment for at least 6 months.
* Minimum age of 18 years old at the screening time
* Reading and comprehension skills of informed consent

Exclusion Criteria:

* Previous retinal treatment for CSC, except for Acetazolamide and Eplerenone
* No diffuse retinal epitheliopathy
* Other concomitant ocular diseases, such as age related macular degeneration, diabetic retinopathy, choroidal neovascularization
* Not controlled glaucoma with eyedrops, or advanced glaucoma
* Myopia or hypermetropia greater than 6 diopters
* Opacities of dioptric media
* Low quality of optical coherence tomography (OCT) and OCT-Angiography scans
* Low quality images of Fluorescein angiography and indocyanine green angiography
* No written consensus signed.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old, with diagnosis of central serous chorioretinopathy since at least 6 months, undergone Acetazolamide and/or Eplerenone therapy with no improvement after 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Vessel density changes | 12 and 24 months
  Evaluation of changes in vessel density of choriocapillaris by optical coherence tomography (OCT) angiography before and after treatment

SECONDARY OUTCOMES:
Choroidal thickness | 12 and 24 months
  Evaluation of changes in choroidal thickness before and after treatment.
Choroidal thickness and vessel density | 12 and 24 months
  Correlation among changes in choroidal thickness and changes in vessel density of choriocapillary with best corrected visual acuity.
Qualitative analysis of retino-choroidal vascularization with identification of vascular pattern | 12 and 24 months
  To qualitatively evaluate the vascular patterns using optical coherence tomography (OCT) - angiography and to verify if a particular one is associated with a greater response to subthreshold micropulse laser treatment.
Metamorphopsia | 12 and 24 months
  Evaluation of quantitative improvement of metamorphosia by M-CHARTS after treatment.
Metamorphopsia and BCVA | 12 and 24 months
  Correlation between metamorphopsia and best corrected visual acuity (BCVA)
Ellipsoid Zone Integrity | 12 and 24 months
  Evaluation of ellipsoid zone integrity by optical coherence tomography (OCT) B scan.
Improvement in retinal function | 12 and 24 months
  To evaluate the potential improvement in retinal function with mean retinal sensitivity and microperimetry.
Quality of life (QoL) | 12 and 24 months
  Evaluation of correlation among quality of life parameters assessed by visual function questionnaire (VFQ), stress and relapses and visual acuity.
Ellipsoid zone and BCVA | 12 and 24 months
  To evaluate the association between ellipsoid zone integrity on optical coherence tomography (OCT) B scan and best corrected visual acuity (BCVA)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli, IRCCS, Roma, R, Italy

IPD SHARING:
Plan to Share IPD: Undecided